CLINICAL TRIAL: NCT04241198
Title: Home Retinal Imaging Using NOTAL-OCT V3.0
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: Home Imaging using NOTAL-OCT
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-04

CONDITIONS: A. AMD Patients, Where at Least One Eye is With Active CNV, Presenting Retinal Fluid at the Enrolment Visit, Undergoing Active Anti-VEGF Treatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will include up to 30 AMD patients, recruited by two medical centers, Tel-Aviv medical center and Assuta Hashalom medical center. At the screening visit, the patients will be imaged in their tested, eligible eye(s), using a commercial Zeiss Cirrus or Heidelberg Spectralis OCT.

DETAILED DESCRIPTION:
Screening visit:

For patients eligible to participate in the study, the following procedure will be done in the "screening visit" at the clinic:

1. Patient will sign the IC (Informed Consent) form
2. The following demographic and clinical data will be collected and registered in the CRF:

   1. Patient's DOB and gender.
   2. Patient's diagnosis in study eye(s), based on patient's medical record, including media opacity (e.g. cataract or corneal opacity, if exists).
   3. Bio-microscopy testing.
   4. Refraction correction by an optometrist.
   5. Habitual Snellen visual acuity
   6. Commercial OCT scanning using Zeiss Cirrus or Heidelberg Spectralis.

OCT scanning pattern:

* Macular cube of at least 6X6mm (20 degrees)
* At least 40 B-scans per cube

Setup and tutorial home visit:

The device will be delivered to the patient's home with a setup guide attached to the package. The patient will read the setup guide instructions, unpack the device, place it on a table and connect it to a power supply. Upon first usage a tutorial clip, explaining how to operate the device and self-image the eyes, will be automatically displayed on the device's external screen. Following the tutorial patients will be instructed to scan their study eye(s). A remote support service, provided by the sponsor, will be available as needed. Its phone number will be given to the patient and will be attached to the device's base.

Daily home testing:

For each eligible eye, the following procedure will be done in the "Daily testing" at the patients' homes:

1. The patients will be requested to self-scan their study eye(s) daily, using the NOTAL-OCT V3.0..
2. The patient will be able call the sponsor's remote support service, during working hours, for assistance in case of questions or problems regarding the operation the NOTAL-OCT V3.0 device.

Exit visit:

For each eligible eye, the following procedure will be done in the "Exit visit" at the clinic:

1. Bio-microscopy testing.
2. Refraction correction by an optometrist.
3. Habitual Snellen visual acuity
4. Commercial OCT scanning using Zeiss Cirrus or Heidelberg Spectralis.

OCT scanning pattern:

* Macular cube of at least 6X6mm (20 degrees)
* At least 40 B-scans per cube NOTAL-OCT V3.0 Scanning.

  6.Patient's experience questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to give informed consent (IC)
2. 18 years of age or older at the time of IC
3. Tested eye(s) diagnosed with AMD
4. Visual acuity of 20/400 Snellen (6/120) or better in the study eye
5. At least one eye is with active CNV, presenting retinal fluid at the enrolment visit, undergoing active anti-VEGF treatment
6. Ability to undergo OCT testing

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AMD patients, where at least one eye is with active CNV, presenting retinal fluid at the enrolment visit, undergoing active anti-VEGF treatment
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
To describe the dynamics of retinal fluid | 30 days
  To describe the dynamics of retinal fluid in eyes undergoing anti-VEGF therapy as manifested in self-operated OCT in daily home testing

SECONDARY OUTCOMES:
To evaluate patient experience when self-operating the Notal-OCT V3.0. | 30 days
  by a patient experience questionnaire.
E. To evaluate the level of agreement between OCT images captured by Notal-OCT V3.0 and a commercial OCT | 30 days
  E. To evaluate the level of agreement between OCT images captured by Notal-OCT V3.0 and a commercial OCT, for the presence of fluid, in the central 10 degrees of the macula, at screening and exit visits.

CONTACTS AND LOCATIONS:
Overall Officials: michaela Glodstein, Dr, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- TLV Medical Center, Tel Aviv, Israel